CLINICAL TRIAL: NCT04331925
Title: Impact of Journal Program on Wellbeing of NICU Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Laura Shashy, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 181831
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Anxiety; Depression
Keywords: NICU parents; Journaling
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety and depression screening (Other): Hospital Anxiety and Depression Scale (HADS) questionnaire administered at the start of the study. After two weeks or at the time of discharge, participants will complete the HADS questionnaire again
  Interventions: Behavioral: Anxiety and depression screening; Behavioral: Journaling
- Anxiety and depression screening with journaling (Experimental): Parents randomized into the intervention group be given verbal instructions to use a journal how/when they choose for the duration of the intervention period. They will also complete the HADS questionnaire before and after the intervention period of two weeks. At the end of the intervention period, these parents will also complete a survey regarding their experience with journaling
  Interventions: Behavioral: Journaling

INTERVENTIONS:
Behavioral: Anxiety and depression screening — At the time of consent, the participant parent will be randomized into either the control or intervention groups. The control group will complete the Hospital Anxiety and Depression Scale (HADS) questionnaire at the start of the study. After two weeks or at the time of discharge, the control group will complete the HADS questionnaire again.
  Arms: Anxiety and depression screening
Behavioral: Journaling — Parents randomized into the intervention group be given verbal instructions to use a journal how/when they choose for the duration of the intervention period

SUMMARY:
The purpose of this study is to investigate the impact of a journaling program on rates of anxiety and depression in neonatal intensive care unit (NICU) parents.

ELIGIBILITY:
Inclusion Criteria:

* Mother, father, and/or legal guardian of infant
* > 28 weeks gestation
* At least 5 days anticipated admission in Vanderbilt NICU

Exclusion Criteria:

* < 28 weeks gestation
* Expected death or discharge within 5 days of admission
* Primary medical team feels that participation would be disruptive or detrimental to infant's care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change in HADS anxiety score | Baseline to 2-4 weeks
  The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. The range of scores for anxiety is 0 to 21. A score of 0 is no anxiety. A score of 1-7 indicates some anxiety. A score of greater than or equal to 8 is the cut-off for clinical anxiety.
Change in HADS depression score | Baseline to 2-4 weeks
  The HADS is a fourteen item scale that generates: Seven of the items relate to depression and seven relate to anxiety. The range of scores for depression is 0 to 21. A score of 0 is no depression. A score of 1-7 indicates some depression. A score of greater than or equal to 8 is the cut-off for clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weitlauf, PHD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Russell LN, Gregory ML, Warren ZE, Weitlauf AS. Uptake and impact of journaling program on wellbeing of NICU parents. J Perinatol. 2021 Aug;41(8):2057-2062. doi: 10.1038/s41372-021-00983-1. Epub 2021 Mar 1. PMID 33649444